CLINICAL TRIAL: NCT03297112
Title: Subharmonic Contrast Ultrasound for Improved Characterization for Adnexal Masses-A Pilot Study
Brief Title: Contrast-Enhanced Subharmonic Ultrasound Imaging in Improving Characterization of Adnexal Masses in Patients Undergoing Surgery
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Lantheus Medical Imaging (Industry)
Responsible Party: Principal Investigator, Flemming Forsberg, Professor - Radiology, Thomas Jefferson University
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16F.394; JT 9149 (Other: JeffTrial Number); R21CA190930 (NIH)
Record Dates: First submitted 2017-09-18; First posted 2017-09-29 (Actual); Results first posted 2019-09-25 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Adnexal Mass
MeSH Terms: interventions — perflutren

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- contrast-enhanced subharmonic ultrasound imaging (Experimental): Patients receive perflutren lipid microspheres IV. After 15 minutes, patients receive perflutren lipid microspheres IV again over 5 minutes and undergo contrast-enhanced subharmonic ultrasound imaging over 60 minutes.
  Interventions: Drug: Perflutren Lipid Microspheres; Procedure: Contrast-Enhanced Subharmonic Ultrasound Imaging

INTERVENTIONS:
Drug: Perflutren Lipid Microspheres — Given IV
  Other Names: Definity
Procedure: Contrast-Enhanced Subharmonic Ultrasound Imaging — Undergo contrast-enhanced subharmonic ultrasound imaging

SUMMARY:
This pilot clinical trial studies how well contrast-enhanced subharmonic ultrasound imaging works in improving the characterization of adnexal masses in patients undergoing surgery. Contrast-enhanced subharmonic ultrasound imaging uses high-frequency sound waves to produce images of internal organs and when combined with an ultrasound agent such as perflutren lipid microspheres, may help improve imaging and management of adnexal masses.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To develop qualitative subharmonic imaging (SHI) or SHI-derived quantitative biomarkers.

II. To generate pilot data for a study to evaluate if they improve the characterization of benign and malignant adnexal masses compared to standard ultrasound or contrast enhanced magnetic resonance imaging (MRI) or the risk of malignancy index (RMI).

SECONDARY OBJECTIVES:

I. To compare the SHI depiction of adnexal masses' neovascularity in humans to intra-tumoral microvascular density (iMVD) obtained from CD31 an immunohistochemical marker of angiogenesis.

ELIGIBILITY:
Inclusion Criteria:

* Be diagnosed with an adnexal mass
* Be scheduled for surgery to remove the adnexal mass
* Be clinically stable
* If a female of child-bearing potential, must have a negative pregnancy test
* Be conscious and able to comply with study procedures
* Have read and signed the Institutional Review Board (IRB)-approved informed consent form for participating in the study

Exclusion Criteria:

* Females who are pregnant or nursing
* Patients who have received an investigational drug in the 30 days before study drug administration, or will receive one within 72 hours (h) afterwards
* Patients with known or suspected right-to-left, bi-directional, or transient right-to-left cardiac shunts
* Patients with pulmonary hypertension or unstable cardiopulmonary conditions
* Patients currently on chemotherapy or with other primary cancers requiring systemic or hepatic loco-regional treatment
* Patients who are clinically unstable, patients who are seriously or terminally ill with a life expectancy of less than 1 month, and patients whose clinical course are unpredictable; for example:

  * Patients on life support or in a critical care unit
  * Patients with unstable occlusive disease (e.g., crescendo angina)
  * Patients with clinically unstable cardiac arrhythmias, such as recurrent ventricular tachycardia
  * Patients with uncontrolled congestive heart failure (New York Heart Association [NYHA] class IV)
  * Patients with recent cerebral hemorrhage
  * Patients who have undergone surgery within 24 hours prior to the study sonographic examination
* Patients with a history of anaphylactic allergy to Definity, manifested by one or more of the following symptoms: generalized urticaria, difficulty in breathing, swelling of the mouth and throat, hypotension, or shock
* Patients with congenital heart defects
* Patients with severe emphysema, pulmonary vasculitis, or a history of pulmonary emboli
* Patients with respiratory distress syndrome
* Patients with thrombosis within the splenic vein

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-09-04 (Actual); Study Completion 2018-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Flemming Forsberg, PhD, Principal Investigator — Sidney Kimmel Cancer Center at Thomas Jefferson University
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Thomas Jefferson University Hospital — http://hospitals.jefferson.edu/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Contrast-enhanced Subharmonic Ultrasound Imaging
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Contrast-enhanced Subharmonic Ultrasound Imaging
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Diagnostic Accuracy of Subharmonic Ultrasound Imaging Compared to Standard Ultrasound or Contrast Enhanced Magnetic Resonance Imaging (MRI)
Description: The techniques will be compared using an analysis of variance (ANOVA) method (i.e., baseline ultrasound imaging, SHI, or MRI) as the dependent variable and outcome as the independent variables. Diagnostic accuracy of lesion identification as "no lesion seen", "definitely benign", "indeterminate" or "definitely malignant" based on independent reads by experience radiologists for SHI with and without contrast vs contrast-enhanced MRI (quantitative analysis). For qualitative analysis, digital images from the SHI imaging were reviewed by the independent radiologists for interpretation. Diagnostic accuracy reported as percentage of lesions correctly identified through SHI as compared to ultrasound or MRI as the gold standard.
Time Frame: Baseline scan to day of surgery
Measure: Number; unit: percent accurate lesion identification
Units Other Than Participants: lesions
Arm/Group | Contrast-enhanced Subharmonic Ultrasound Imaging
Number analyzed (Participants) | 12
Number analyzed (lesions) | 12
percent accurate lesion identification
  Qualitative analysis of CEUS SHI with contrast | 70
  Qualitative analysis of CEUS SHI without contrast | 56

2. Primary Outcome: Accuracy of SHI Characterization Compared to the Risk of Malignancy Index
Description: The ability of SHI to accurately characterize lesions as benign from malignant masses as compared to other imaging (ultrasound or MRI) and pathology will be analyzed using logistic regression and receiver operating characteristic (ROC) analyses.
Time Frame: Baseline scan to day of surgery
Measure: Number; unit: percent accurate m lesion identification
Arm/Group | Contrast-enhanced Subharmonic Ultrasound Imaging
Number analyzed (Participants) | 12
percent accurate m lesion identification | 73

ADVERSE EVENTS:
Time Frame: 30 minutes after the second Definity injection
Arm/Group | Contrast-enhanced Subharmonic Ultrasound Imaging
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-12): https://cdn.clinicaltrials.gov/large-docs/12/NCT03297112/Prot_SAP_000.pdf